CLINICAL TRIAL: NCT06976723
Title: The Effect of Treatment Onset Time on Acute Treatment Efficacy in Migraine Patients Using Remote Electrical Neuromodulation (REN)
Brief Title: Nerivio Efficacy by Time of Treatment Onset
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Theranica (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RWE-010
Record Dates: First submitted 2025-04-24; First posted 2025-05-16 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-05

CONDITIONS: Migraine; Acute Treatment of Migraine
Keywords: Nerivio; Remote Electrical Neuromodulation
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: 1. - Nerivio treatments within 60 minutes from migraine attack onset
  2. - Nerivio treatments over 60 minutes from migraine attack onset
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Early treatment (Active Comparator): Nerivio treatment was administered within 60 minutes of migraine onset
  Interventions: Device: Nerivio
- Late treatment (Active Comparator): Nerivio treatment was administered more than 60 minutes after migraine onset
  Interventions: Device: Nerivio

INTERVENTIONS:
Device: Nerivio — Remote electrical neuromodulation (REN) device for the acute treatment of migraines. The device delivers transcutaneous electrical stimulation to the upper arm to induce conditioned pain modulation (CPM) that activates a descending endogenous analgesic mechanism. The treatment is self-administered and controlled by a smartphone application

SUMMARY:
This is a Post-marketing study investigating the impact of treatment time onset with Nerivio on the efficacy of Remote Electrical Neuromodulation (REN) for the acute treatment of migraine.

Efficacy will be evaluated as a change in headache pain severity and functional disability from baseline to 2 hours post-treatment in at least 50% of the treatments, based on the treatment start time from the beginning of the migraine attack.

DETAILED DESCRIPTION:
The REN device (Nerivio by Theranica, ISRAEL) is a neuromodulation device approved by the FDA for acute and/or preventive treatment of migraine in patients 8 years old and above. It is a wearable device applied to the upper arm. It stimulates C and Aδ noxious fibers using a modulated, symmetrical, biphasic, square pulse with a pulse width of 400 μs, modulated frequency of 100-120 Hz, and up to 40 mA output current, which the patient can adjust. The REN device is operated by a designated app that is downloaded to the user's phone prior to first use of the Nerivio device. As part of the sign-up process for the Nerivio app, all patients accept the terms of use, which specify that providing personal information is done on their own free will and that their de-identified data may be used for research purposes. Users are not obligated to provide personal information and could treat without providing any feedback.

The app includes a secure, personal migraine diary, which enables patients to record and track their migraines and other headaches. At the beginning of each treatment, and again at 2 hours after the start of treatment, patients are prompted to record their symptoms, including pain level (none, mild, moderate, severe), functional disability (None, Mild limitation, Moderate limitation, Severe limitation), and an indication of which medications, if any, were taken within that 2-hour time window.

Post-marketing surveillance is designed to assess the safety, utilization, and efficacy in larger and more diverse populations and in various real-world environments and situations. As a digital therapeutic device (i.e., electroceutical), the REN device enables prospective collection of electronic patient-reported outcomes in real-world clinical practice. This post-marketing RWE study investigates the impact of early treatment (within 60 minutes from the migraine onset) vs. late treatment (over 60 minutes from the migraine onset) on the effectiveness of the Nerivio treatment of acute migraine.

for this study, treatments were classified as 'early treatments' if Nerivcio was administered within 1-hour (60 minutes) of migraine onset and classified as 'late treatments' if administered more than 1-hour (60 minutes) after onset. On a patient level, a patient was defined as an 'early-treater' if s/he had reported treatment onset in at least two treatments and had treated early in 50% or more of treatments. A patient was defined as a 'late-treater' if s/he had reported treatment onset in at least two treatments and had treated late in more than 50% of treatments.

The following efficacy outcome will be assessed - Pain Relief, Pain Freedom, Functional Disability Relief, Functional Disability Freedom, Freedom from each migraine-associated symptom (Photophobia, Phonophobia, Nausea/Vomiting) and Consistent Efficacy.

ELIGIBILITY:
Inclusion Criteria:

* • Users who had reported treatment onset time in at least one treatment through the REN companion smartphone app

Exclusion Criteria:

* • Treatments that included medications for acute treatment of migraine

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55261 (Actual)
Dates: Start 2025-05-07 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Pain Relief | 2 hours post treatment
  Proportion of treatments in which there was a reduction in headache intensity from moderate or severe headache at baseline to mild or no pain 2 hours post-treatment.
Pain Freedom: | 2 hours post treatment
  Proportion of treatments in which there was a reduction in headache intensity from mild or moderate or severe headache at baseline to no headache 2 hours post-treatment.

SECONDARY OUTCOMES:
Functional Disability Relief | 2 hours post treatment
  Proportion of treatments in which there was at least one-grade improvement in functional disability level at baseline to 2 hours post-treatment.
Functional Disability Freedom | 2 hours post treatment
  Proportion of treatments in which there was a reduction in functional disability level at baseline to no functioal disability at 2 hours post-treatment.
Freedom from each migraine-associated symptom (Photophobia, Phonophobia, Nausea/Vomiting) | 2 hours post treatment
  Proportion of treatments in which there was an absence of each of the three associated symptoms 2 hours post-treatment in treatments with reported associated symptoms at baseline
Consistent efficacy | 2 hours post treatment
  The proportion of responders in each of the efficacy outcomes at 2 hours post treatment. A responder is defined as a subject who presented efficacy in at least 50% of their treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Alit Stark-Inbar, PhD, Principal Investigator — Theranica
Locations (1):
- Theranica Bio-Electronics Inc, Bridgewater, New Jersey, United States